CLINICAL TRIAL: NCT06337448
Title: Light Emitting Diode in the Treatment of Vulvodynia: a Pilot Study
Brief Title: Light Emitting Diode in the Treatment of Vulvodynia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Principal Investigator, Patricia Lordelo, Head of the CentroAAP, Centro de Atenção ao Assoalho Pélvico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74090923.9.0000.5544
Record Dates: First submitted 2024-03-04; First posted 2024-03-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Vulvodynia
Keywords: vulvodynia; Light-emitting diode
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Light-emitting diode (Experimental): The LED application protocol will be carried out with external use equipment model Antares, from the company IBRAMED (Amparo, São Paulo, Brazil), with a cluster G2 applicator. The power will be 450mW/cm2 and dose 5J/cm2 for 2 minutes and 13 seconds (automatic programming) in 450nm waves (blue wavelength). The treatment consists of eight sessions, carried out daily, except on weekends. The patient will remain naked, in a closed room, in the lithotomy position on a gynecological table, in the presence of only a physiotherapist specializing in women's health, who will apply the light.
  Interventions: Device: Blue LED

INTERVENTIONS:
Device: Blue LED — The patient will remain naked, in a closed room, in the lithotomy position on a gynecological table, and he LED will be positioned in the direction of the patient's genitalia, keeping the internal and external vulvar lips open, so the LED can reach the largest possible region for therapeutic action.

SUMMARY:
Vulvar pain can be related to a specific cause (inflammation, cancer, trauma, infection) or can be classified as vulvodynia, when vulvar pain is idiopathic and lasts for at least three months. The main symptoms reported are pain, burning, erythema, increased sensitivity, itching and burning, which affect the quality of life, psycho-emotional well-being, relationships and sexual function of these women. Photobiomodulation has been described in the literature as an alternative to treat pain. Our group has studied blue LED for some vulvovaginal dysfunctions and, due to the positive sensory effects observed in patients with vaginal stenosis and genitourinary syndrome of menopause, it is hypothesized that this technique could also bring beneficial effects for women with vulvodynia. A pilot study will be carried out, with descriptive data, with 10 women with vulvodynia. Participants will be evaluated with a basic anamnestic questionnaire and sociodemographic data. The following questionnaires will be used: Female Sexual Function Index (FSFI), Sexual Quotient - Female Version, Vulvar Pain Assessment Questionnaire. After answering the questionnaires, the volunteer will undergo a perineal physical assessment by an experienced physiotherapist, which includes a) inspection of the genital region, reflex tests, assessment of the functions of the pelvic floor muscles, b) the cotton swab test to evaluate painful sensitivity in the vestibule, c) the tampon test to evaluate painful sensitivity in the introitus and vaginal canal. Pain assessments will be quantified by the visual analogue pain scale (VAS), which ranges from 0 (no pain) to 10 (maximum pain). At the end of the treatment, the participant will answer the questionnaires again, undergo reassessment of pain sensitivity in vulva, introitus and vaginal canal, of the function of the pelvic floor muscles and will be asked "What is your perception of improvement" and "What is your level of satisfaction with the treatment?". The answers will be giving according to a Likert Scale of five points. The LED application protocol will be carried out with external use equipment model Antares, from the company IBRAMED (Amparo, São Paulo, Brazil), with a cluster G2 applicator. The power will be 450mW/cm2 and dose 5J/cm2 for 2 minutes and 13 seconds (automatic programming) in 450nm waves (blue wavelength). The treatment consists of eight sessions, carried out daily, except on weekends.

ELIGIBILITY:
Inclusion Criteria:

* vulvodynia diagnosis

Exclusion Criteria:

* patients diagnosed with vaginal infection
* difficulty in understanding the proposed instruments
* patients with chronic degenerative neurological diseases
* pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-16 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Visual Analogue Scale. | During the all 8 sessions (daily), at the end (one week after de beginning of the treatment) and one month after the end of the treatment.
  To assess the safety of the treatment regarding the genital's sensation (burning, itching, pain) and genital's visual aspects (lesion, erosion, redness).
Tolerability of participants to the treatment assessed by Likert Scale. | During the all 8 sessions (daily) and at the end (one week after de beginning of the treatment).
  To assess the tolerability of the patient according to the Likert 5 Points Scale: very comfortable, comfortable, nor comfortable nor discomfortable, discomfortable, impossible to tolerate the treatment.
Evaluate the clinical response assessed by the Visual Analogue Scale. | At the beginning of the treatment and at the end (one week after de beginning of the treatment), 1, 3 and 6 months after the end treatment.
  To assess the clinical effect of the treatment it will be used the Visual Analogue Scale (VAS), which varies from 0 to 10. The pain will be assessed on the swab test and the tampon test in the genital area. Minimum decrease in 2 points on the VAS will be interpretated as clinical effect.
Evaluate the clinical response assessed by a questionnaire. | At the beginning of the treatment and at the end (one week after de beginning of the treatment), 1, 3 and 6 months after the end treatment.
  To assess the clinical effect of the treatment it will be used the Vulvar Pain Assessment Questionnaire: the higher the score, the greater the intensity of pain and impairment of the assessed domains.

SECONDARY OUTCOMES:
Evaluate the sexual function of women with vulvodynia by Female Sexual Function Index (FSFI). | At the beginning of the treatment and at the end (one week after de beginning of the treatment), 1, 3 and 6 months after the end of the treatment.
  The FSFI has 19 items, the score varies from 2 to 36, and the cut-off point is 26, meaning that scores of 26 or less classify the patient as having sexual dysfunction.
Evaluate the sexual function of women with vulvodynia by Sexual Quotient - Female Version (SQ-FV). | At the beginning of the treatment and at the end (one week after de beginning of the treatment), 1, 3 and 6 months after the end treatment.
  The FQ-SV has 10 items and the score varies from 0 to 100. Higher values indicate better sexual performance/satisfaction. The score classification is 82-100 points: good to excellent; 62-80 points: regular to good; 42-60 points: unfavorable to fair; 22-40 points: poor to unfavorable; 0-20 points: nil to bad. A cutoff point of 60 (between 48 and 84) was established as a means of screening for female sexual dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao assoalho pélvico, Salvador, Estado de Bahia, Brazil